CLINICAL TRIAL: NCT03694470
Title: Retrospective Study to Describe Characteristics of Patients With Type 2 Diabetes Mellitus Who Were Initiating Use or Treatment With Sodium-glucose Co-transporter-2 Inhibitors and Other Diabetes Medications (Other Glucose Lowering Drugs) in 2015-17 Based on National Russian Diabetes Registry Data
Brief Title: Characteristics of Patients With Type 2 Diabetes Mellitus (CVD-RNDR)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00048
Record Dates: First submitted 2018-09-03; First posted 2018-10-03 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational retrospective study will describe characteristics of patients with type 2 diabetes mellitus (T2DM) who were initiating use or treatment with sodium-glucose co-transporter-2 (SGLT-2) inhibitors and other diabetes medications (other glucose lowering drugs) in 2015-17 based on National Russian Diabetes Registry data.

ELIGIBILITY:
Inclusion criteria are:

* New user receiving or dispensed prescription of SGLT-2 inhibitor medication or other GLD treatments oral as well as injectable, including fixed-dose combination (FDC) products containing these medication groups;
* T2DM diagnosis on or prior to the index year;
* ≥ 18 years old at index year.

Exclusion criteria are:

* Patients with a T1DM diagnosis on or prior to index year and only insulin use in the year prior to index;
* Patients with a gestational diabetes in the index year or 1 year prior to index.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data of T2DM patients consecutively included in the RNDR from January 2015 to October 2017 will be included in this retrospective analysis. New users will be defined as individuals with T2DM either receiving a prescription of a SGLT-2 inhibitor or other GLD during the study period. Individuals with a previous issued/dispensed prescription of that medicine class during the preceding 1 year are not defined as new users. The year of the first issued prescription of the included medication classes during the study period will be denoted the index year. The group of other GLD will include all diabetes medicines, allowing combinations and monotherapy use except use of SGLT-2 inhibitors. The class SGLT-2 inhibitors include mainly dapagliflozin, empagliflozin and canagliflozin.
  Since SGLT-2 inhibitors are relatively recently introduced on the market the population size and follow-up time is limited. Approximately 22,000 patients registered in RNDR will be included.
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who were new users of SGLT-2 inhibitors in 2015, 2016, 2017 | 2015-2017
  The proportion of patients who were new users of SGLT-2 inhibitors in 2015, 2016 2017 among T2DM patients initiated use of antidiabetic treatment in these years according to Russian National Diabetes Registry data.

SECONDARY OUTCOMES:
Number of participants with abdominal laboratory values | 2015-2017
  Number of participants with abdominal laboratory values glycosylated haemoglobin (Hb1Ac), total Cholesterol, low Density Lipids (LDL), high Density Lipids (HDL), creatinine, estimated Glomerular Filtration Rate (EGFR)
Number of participants with co-morbidities | 2015-2017
  Number of participants with co-morbidities: myocardial infarction (MI), stroke (ischemic or hemorrhagic )Transient Ischemic Attack (TIA)Peripheral Artery Disease (PAD), Heart Failure, Hypertension, Hyperlipidemia, Neuropathy, Nephropathy, Retinopathy, Therapies, Diabetes medications, Hypertension medications, Diuretics, Lipid lowering drugs, Anti-platelets.

CONTACTS AND LOCATIONS:
Locations (1):
- Research site, Moscow, Russia

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=34929&filename=D1690R00048_Study_report_synopsis.pdf